CLINICAL TRIAL: NCT04363853
Title: Treatment of Serious and Critical Patients With COVID-19 With Tocilizumab
Brief Title: Tocilizumab Treatment in Patients With COVID-19
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, MD MSc Head of Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INF-3343-20-22-1
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Phase II, single-arm, open-label, prospective, blinded, clinical trial with Tocilizumab as the sole agent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tocilizumab tratment (Experimental): Tocilizumab (RoActembra). Vials of 20 ml with 400 mg (20mg/ml) and 4ml with 80 mg (20mg/ml). A singe 60-minute IV infusion of 8mg/kg (maximum dose of 800 mg). Dose was not adjusted for weight more than 100 kg. After first dose, if fiver persists within 12 hours, a second dose was administrated.
  A maximum of two doses was allowed.
  Interventions: Drug: Tocilizumab 20 MG/ML

INTERVENTIONS:
Drug: Tocilizumab 20 MG/ML — We study the impact of the administration of Tocilizumab on the evolution of the acute respiratory distress syndrome (ARDS) in patients with severe or critical SARS-CoV-2 infection.

SUMMARY:
A phase II clinical trial will be carried out with the objective of studying the impact of the administration of Tocilizumab on the evolution of the acute respiratory distress syndrome (ARDS) in patients with severe or critical SARS-CoV-2 infection. Due to the high mortality of severe forms of SARS-CoV-2 and for ethical reasons, a control arm will not be included. Patients will be recruited by signing an informed consent and the baseline variables of interest will be recorded. Tocilizumab will be administered in one or two doses, depending on the case, and will be followed up for 30 days. The response to treatment, survival and evolution will be studied. Factors associated with improvement of ARDS and survival will be identified through multivariate analyzes. The results will be compared with those reported internationally.

DETAILED DESCRIPTION:
In December 2019, a group of patients with the acute respiratory disease was detected in Wuhan, Hubei Province of China. A month later, a new beta-coronavirus was identified as the cause of the 2019 coronavirus infection. Despite China's efforts to contain the disease, it spread rapidly outside the continent. Currently, Mexico is one of the countries that is facing this world health problem with a dynamic and exponential increase in the number of confirmed cases.

SARS-CoV-2 is a coronavirus that belongs to the group of β-coronaviruses of the subgenus Coronaviridae. The SARS-CoV-2 is the third known zoonotic coronavirus disease after severe acute respiratory syndrome (SARS) and Middle Eastern respiratory syndrome (MERS). The diagnosis of SARS-CoV-2 recommended by the WHO, CDC is the collection of a sample from the upper respiratory tract (nasal and oropharyngeal exudate) or from the lower respiratory tract such as expectoration of endotracheal aspirate and bronchioloalveolar lavage and its analysis using the test of real-time polymerase chain reaction (qRT-PCR).

The clinical manifestations of the patients are heterogeneous presenting asymptomatic symptoms, mild respiratory disease, severe pneumonia, acute respiratory failure syndrome (ARDS), and even death. According to the Berlin definition, ARDS is an acute lung injury that occurs within 7 days after the triggering event and is characterized by bilateral lung infiltrates and severe progressive hypoxemia, as well as non-cardiogenic pulmonary edema. The mortality associated with ARDS depends on its severity: mild 27%, moderate 32%, and severe 45%. In patients with SARS and SARS-CoV-2, the average duration of mechanical ventilation was reported in 10 (7-12) days, achieving extubation in 6/18 (33%) of which their meantime under mechanical ventilation was 11 (7-12) days. Of these patients, none received treatment with tocilizumab, only 1 patient received hydroxychloroquine, and another patient was treated with lopinavir-ritonavir. Therefore, the present study proposes that the use of Tocilizamab will shorten the time to improve, so an evaluation of the ARDS will be carried out at 7 days.

Initial reports suggest that SARS-CoV-2 is associated with a severe illness that requires the intensive care unit in approximately 5% of confirmed infections. In the CDC report from China, the clinical manifestations of the disease were divided into:

Mild: Mild respiratory symptoms (cough, malaise, temperature> 37.5, runny nose) with or without pneumonia data by an imaging study (up to 81% cases) Severe: dyspnea, increase in respiratory rate ≥ 30 breaths / min, oxygen saturation ≤ 93%, PaO2 / FiO2 <300 mmHg, and image lung infiltrates> 50% within 24 to 48 hours of symptom onset (up to 14 % of the cases) Critical: respiratory failure, septic shock and/or multiple organ failure (up to 5% of cases)

China's mortality rate from SARS-CoV-2 was 2.84%, with a ratio of male to female deaths of 3.25: 1. The average age of death was 75 years, and the average time from the first symptom to death was 14 days. For people age 70 and older, the average time from first symptoms to death was shorter than for people younger than age 70. In another retrospective study of 99 cases, 17% of patients developed Acute Respiratory Failure Syndrome (ARDS), and 11% worsened in a few days and died. Critical case mortality has been documented to reach 60.5%, however, Mexico still does not exist epidemiological data because is not yet reached the zenith of the pandemic.

The SARS-CoV-2 infection causes dysregulation of the immune response mediated by cytokines and chemokines. An increase in inflammation-related cytokines including IL-2, IL-7, and IL-10, colony-stimulating factor (G-CSF), protein 10 inducible interferon g (IP10), protein, was reported in plasma samples from patients. monocyte chemoattractant (MCP1), macrophage inflammatory protein 1 alpha (MIP1A), and tumor necrosis factor-alpha (TNF-a), especially in severe patients. This suggests that SARS-CoV-2 patients have a large infiltrate of inflammatory immune cells and severe lung inflammation. IL-6 and IL-10 expression levels increase the risk of progression to a critical condition.

Cytokine storm syndrome is a phenomenon during which there is an immune dysregulation due to the increase of proinflammatory cytokines in response to stimulation by microorganisms or drugs.

Under homeostasis conditions, the body's pro-inflammatory and anti-inflammatory cytokine concentrations remain relatively balanced. Before infection, there may be abnormal and dysregulated activation of dendritic cells, macrophages, lymphocytes, and NK cells. The release and action of a large number of proinflammatory cytokines facilitate a positive feedback loop. After a certain threshold, there may be a cytokine storm. Patients will present with fever, diffuse intravascular coagulation (DIC), shock, and organ failure. The transition from mild to severe disease in COVID-19 patients may be caused by a cytokine storm.

Manifestations of a dysregulated inflammatory response have been identified in patients with COVID-19. The cardinal features of this syndrome include constant fever, cytopenias, and hyperferritinemia. Pulmonary involvement, including ARDS, occurs in approximately 50% of patients. A cytokine profile that resembles LHHS has been associated with COVID-19 disease severity.

At the time of infection, immune mechanisms are activated, including specific and non-specific immune responses. Endogenous viral protein synthesized within infected cells can activate virus-specific CD8 + T cells through the major pathway of the histocompatibility complex-I (MHC-I). There is then proliferation, differentiation, and effector responses of CD8 + T cells (24). Increased IL-2, IL-7, granulocyte colony-stimulating factor, interferon-γ inducible protein 10, monocyte chemoattractant protein 1, macrophage inflammatory protein 1-α, and necrosis factor have been observed in severe cases tumor-α. Continuous and dysregulated amplification exacerbates the manifestations associated with infection, while hypoxia and necrosis eventually lead to an uncontrolled inflammatory response and will trigger cytokine storms. There is a probability that immunosuppression is beneficial in a hyper-inflammatory state.

Therapeutic options include steroids, intravenous immunoglobulin, selective cytokine blockade (eg, Anakinra or Tocilizumab), JAK inhibition, vaccines, reinfusion of serum from recovered patients, progenitor therapy, elimination of immune cells (eg. , Alendizumab, Rituximab), among others.

All patients with severe COVID - 19 should undergo tests for hyper inflammation using laboratory tests such as ferritin levels, platelet count, globulin sedimentation rate, and H score measurement in order to determine the subgroup of patients to whom the immunosuppression may improve the risk of mortality.

A study carried out to identify the immune characteristics of those infected with SARS-CoV-2 showed that patients in the intensive care unit had a significant decrease in hemoglobin and albumin, with an increase in concentrations of the c-reactive protein (PCR), alanine aminotransfer (ALT), aspartate aminotransferase (AST) and lactate dehydrogenase (DHL). The total number of leukocytes did not show significant differences, while the number of lymphocytes decreased significantly. Furthermore, they found an increase in the number of G-CSF and in IL-6, suggesting a high risk of monocyte-mediated release of inflammatory cytokines that can migrate to the lung and produce severe clinical manifestations and even death.

The management of the critically ill adult patient with SARS-CoV-2 is not standardizing, however, the panel of experts from the "Surviving Sepsis Campaign" has published 54 recommendations for the management of the patient with severe SARS-CoV-2 and ARDS. The recommendations focus on hemodynamic support, fluid therapy, use of vasoactive agents, invasive mechanical ventilation, as well as management of the "cytokine storm" syndrome.

One of the proposals for the treatment of cytokine storm and macrophage activation in severe or critical stages of SARS-CoV-2 is the use of drugs that inhibit the interaction of IL-6 with its receptor. Tocilizumab (TCZ) is a humanized recombinant monoclonal antibody of the IgG1 immunoglobulin subclass, is directed against soluble or membrane IL-6 receptors (IL-6R). TCZ inhibits the binding of IL-6 to its receptor by reducing pro-inflammatory activity.

The use of TCZ in patients with severe/critical SARS-CoV-2 was first reported in China. Patients received TCZ treatment at an initial dose of 400 mg with an additional dose in the patient with persistent fever (maximum of two doses). The patients presented a rapid reduction in fever and in the supplemental oxygen requirement in the days after receiving the medication. Despite the promising results of this study, there is currently no solid evidence demonstrating the safety and efficacy of TCZ for the clinical treatment of SARS-CoV-2 pneumonia. The FDA recently approved a randomized, double-blind, placebo-controlled phase III clinical trial to evaluate the safety and efficacy of TCZ (ActemraMR) added to standard care in hospitalized adult patients with severe SARS-CoV-2 disease, which will be held in the United States of America (ClinicalTrials.gov Identifier: NCT04320615). Likewise, Italy is recruiting patients for a phase II study with a single TCZ treatment arm in critically ill patients (ClinicalTrials.gov Identifier: NCT04317092, NCT04315480). China is conducting a study with Tocilizumab vs. renal replacement therapy for the management of cytokine release syndrome (ClinicalTrials.gov Identifier: NCT04306705). In patients with mild-moderate SARS-CoV-2, the US will initiate a phase 2 study in 50 patients to assess its efficacy (ClinicalTrials.gov Identifier: NCT04331795). As well as its comparison with other medications (hydroxychloroquine and azithromycin, ClinicalTrials.gov Identifier: NCT04332094) and combinations (Favipiravir + Tocilizumab vs Favipiravir and Tocilizumab ClinicalTrials.gov Identifier: NCT04310228).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Diagnosis of SARS-CoV-2 infection by RT-PCR
* Diagnosis of serious or critical illness, without mechanical ventilation or with less than 24 hours of mechanical ventilation.
* Severe: dyspnea, increase in respiratory rate ≥ 30 breaths / min, oxygen saturation <90% or PaO2 <60 mmHg or increase in supplemental oxygen requirement more than 3% from baseline, PaO2 / FiO2 <300 mmHg, and / or pulmonary infiltrates by image> 50% within 24 to 48 hours of symptom onset.
* Critical: respiratory failure (alteration in gas exchange with PaO2 <60 mmHg with or without elevation of PaCO2> 33 mmHg), septic shock (hypotension secondary to sepsis with a requirement for vasopressors to maintain a mean arterial pressure> 65 mmHg and lactate> 2 mmol / l).
* Signature of informed consent by the patient, family member or legal representative
* Negative pregnancy test for women of childbearing age.
* Male patients who agree to use barrier methods when having sexual intercourse in the following 80 days after receiving tocilizumab
* Patients receiving immunomodulatory treatment (cancer, transplant recipients or other diseases) that may temporarily suspend the drug.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients who by indication of their treating doctor cannot suspend previous immunomodulatory treatment.
* Known allergic reactions to Tocilizumab or any excipients.
* Patients receiving systemic steroids at a dose greater than 1 mg / Kg of weight per day in prednisone equivalents
* Patients with SOFA score> 15 points that predicts 90% mortality on admission
* The decision of the attending physician not to include the patient due to the presence of any condition that does not allow the administration of the drug to be safe.
* Diverticulitis or intestinal perforation
* Patients with any of the following active infections: viral hepatitis, tuberculosis, HIV infection, bacterial and/or fungal and/or viral infections (other than SARS-CoV-2 infection) suspected or diagnosed using compatible microbiological isolation.
* Alanine aminotransferase/aspartate aminotransferase values> 5 times the upper limit of normal
* Neutrophil values <1000/ml,
* Platelet values <50,000/ml.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematic biometry | 24 hours
  Until removal of mechanical ventilation, Control of hemoglobin, hematocrit, platelet , and leukocytes levels.
Blood chemistry | 24 hours
  Until removal of mechanical ventilation. Control of glucose, uric acid, cholesterol, urea, triglycerides, and creatinine.
Blood gas | 24 hours
  Until removal of mechanical ventilation. Control metabolic and repiratory alcalosis or acidosis.
Hematic biometry | 48 hours
  Until removal of mechanical ventilation, Control of hemoglobin, hematocrit, platelet , and leukocytes levels.
Blood chemistry | 48 hours
  Until removal of mechanical ventilation. Control of glucose, uric acid, cholesterol, urea, triglycerides, and creatinine.
blood gas | 48 hours
  Until removal of mechanical ventilation. Control metabolic and repiratory alcalosis or acidosis.
Hematic biometry | 72 hours
  Until removal of mechanical ventilation, Control of hemoglobin, hematocrit, platelet , and leukocytes levels.
Blood chemistry | 72 hours
  Until removal of mechanical ventilation. Control of glucose, uric acid, cholesterol, urea, triglycerides, and creatinine.
blood gas | 72 hours
  Until removal of mechanical ventilation. Control metabolic and repiratory alcalosis or acidosis.
Hematic biometry | 7 days
  Until removal of mechanical ventilation, Control of hemoglobin, hematocrit, platelet , and leukocytes levels.
Blood chemistry | 7 days
  Until removal of mechanical ventilation. Control of glucose, uric acid, cholesterol, urea, triglycerides, and creatinine.
blood gas | 7 days
  Until removal of mechanical ventilation. Control metabolic and repiratory alcalosis or acidosis.
Hematic biometry | 14 days
  Until removal of mechanical ventilation, Control of hemoglobin, hematocrit, platelet , and leukocytes levels.
Blood chemistry | 14 days
  Until removal of mechanical ventilation. Control of glucose, uric acid, cholesterol, urea, triglycerides, and creatinine.
blood gas | 14 days
  Until removal of mechanical ventilation. Control metabolic and repiratory alcalosis or acidosis.
thorax radiography | 24 hours
  Until removal of mechanical ventilation. Monitoring for signs of pneumonia imaging.
thorax radiography | 7 days
  Until removal of mechanical ventilation. Monitoring for signs of pneumonia imaging.
thorax radiography | 14 days
  Until removal of mechanical ventilation. Monitoring for signs of pneumonia imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Óscar Arrieta, M.D.,M.Sc., Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available in July 2020

REFERENCES:
- [Background] Hui DS, I Azhar E, Madani TA, Ntoumi F, Kock R, Dar O, Ippolito G, Mchugh TD, Memish ZA, Drosten C, Zumla A, Petersen E. The continuing 2019-nCoV epidemic threat of novel coronaviruses to global health - The latest 2019 novel coronavirus outbreak in Wuhan, China. Int J Infect Dis. 2020 Feb;91:264-266. doi: 10.1016/j.ijid.2020.01.009. Epub 2020 Jan 14. No abstract available. PMID 31953166
- [Background] Paules CI, Marston HD, Fauci AS. Coronavirus Infections-More Than Just the Common Cold. JAMA. 2020 Feb 25;323(8):707-708. doi: 10.1001/jama.2020.0757. No abstract available. PMID 31971553
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Hu X, Deng Y, Wang J, Li H, Li M, Lu Z. Short term outcome and risk factors for mortality in adults with critical severe acute respiratory syndrome (SARS). J Huazhong Univ Sci Technolog Med Sci. 2004;24(5):514-7. doi: 10.1007/BF02831124. PMID 15641708
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Lu H, Stratton CW, Tang YW. Outbreak of pneumonia of unknown etiology in Wuhan, China: The mystery and the miracle. J Med Virol. 2020 Apr;92(4):401-402. doi: 10.1002/jmv.25678. Epub 2020 Feb 12. No abstract available. PMID 31950516
- [Background] Schmitt J, Boutonnet M, Goutorbe P, Raynaud L, Carfantan C, Luft A, Pasquier P, Meaudre E, Bordes J. Acute respiratory distress syndrome in the forward environment. Retrospective analysis of acute respiratory distress syndrome cases among French Army war casualties. J Trauma Acute Care Surg. 2020 Aug;89(2S Suppl 2):S207-S212. doi: 10.1097/TA.0000000000002633. PMID 32102034
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Wang W, Tang J, Wei F. Updated understanding of the outbreak of 2019 novel coronavirus (2019-nCoV) in Wuhan, China. J Med Virol. 2020 Apr;92(4):441-447. doi: 10.1002/jmv.25689. Epub 2020 Feb 12. PMID 31994742
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096